CLINICAL TRIAL: NCT00749541
Title: 25 Hydroxy Vitamin d Levels in Patients Undergoing an Elective Coronary Catheterization
Brief Title: Vitamin d Levels and Coronary Catheterization
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: dr. renana shor, assaf harofeh medical center internal medicine a
Other Study IDs: vitamin d
Record Dates: First submitted 2008-09-07; First posted 2008-09-09 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2008-09

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin d coronary catheterization
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1normal catheter.
- abnormal catheter.

SUMMARY:
decreased vitamin d levels are associated with increased inflammatory markers,and renin angiotensin levels.

decreased levels were also found to be connected to increased cardiovascular mortality.

we therefore hypothesise that in patients with pathological results of coronary catheterization we will find decreased levels of 25 hydroxy vitamin d.

we will examine patients undergoing elective coronary catheterization and compare two groups: those with normal results and those with pathological results.

ELIGIBILITY:
Inclusion Criteria:age

* >18 years,
* no known ihd

Exclusion Criteria:

* renal failure ,
* medications including vitamin d, calcium ,phosphate
* hyper or hypoparathyroidism,
* abnormal calcium or phosphate values,
* known pathological coronary catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing an elective coronary catheterization over the age of 18.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: renana shor, md, Principal Investigator — assaf harofeh mc
Locations (1):
- Assaf Harofeh Mc, Ẕerifin, Israel